CLINICAL TRIAL: NCT01626378
Title: A Double-Blind, Placebo-Controlled, Randomized, Parallel Group, 12-Month Safety and Efficacy Trial of TRx0237 in Subjects With Behavioral Variant Frontotemporal Dementia (bvFTD)
Brief Title: Safety and Efficacy Study Evaluating TRx0237 in Subjects With Behavioral Variant Frontotemporal Dementia (bvFTD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TauRx Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRx-237-007
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Behavioral Variant Frontotemporal Dementia (bvFTD)
Keywords: Behavioral Variant Frontotemporal Dementia; bvFTD; Frontotemporal Dementia
MeSH Terms: conditions — Frontotemporal Dementia | interventions — hydromethylthionine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TRx0237 200 mg/day group (Experimental)
  Interventions: Drug: TRx0237
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRx0237 — TRx0237 100 mg tablet will be administered twice daily.
  Arms: TRx0237 200 mg/day group
Drug: Placebo — Placebo tablets will be administered twice daily. The placebo tablets include 4 mg of TRx0237 as a urinary and fecal colorant to maintain blinding; hence, the placebo group will receive a total of 8 mg/day of TRx0237.
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the safety and efficacy of TRx0237 in the treatment of patients with behavioral variant frontotemporal dementia (bvFTD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable bvFTD
* Centrally rated frontotemporal atrophy score of 2 or greater on brain MRI
* MMSE ≥20
* Age <80 years
* Modified Hachinski ischemic score of ≤ 4
* Females, if of child-bearing potential, must practice true abstinence or be competent to use adequate contraception and agree to maintain this throughout the study
* Subject, and/or, in the case of reduced decision-making capacity, legally acceptable representative(s) consistent with national law is/are able to read, understand, and provide written informed consent
* Has one (or more) identified adult caregiver who is willing to provide written informed consent for his/her own participation; is able to read, understand, and speak the designated language at the study site; either lives with the subject or sees the subject for ≥2 hours/day ≥3 days/week; agrees to accompany the subject to each study visit; and is able to verify daily compliance with study drug
* If currently taking an acetylcholinesterase inhibitor and/or memantine, the subject must have been taking such medication(s) for ≥3 months. The dosage regimen must have remained stable for ≥6 weeks and it must be planned to remain stable throughout participation in the study.
* Able to comply with the study procedures

Exclusion Criteria:

* Significant central nervous system (CNS) disorder other than bvFTD
* Significant intracranial pathology seen on brain MRI scan
* Biomarker evidence of underlying Alzheimer's disease pathology
* Expressive language deficits
* Meets research criteria for Amyotrophic Lateral Sclerosis or motor neuron disease
* Meets diagnostic criteria for probable bvFTD but has a proven mutation producing non-tau, non-TDP-43 pathology
* Clinical evidence or history of stroke, transient ischemic attack, significant head injury or other unexplained or recurrent loss of consciousness ≥15 minutes
* Epilepsy
* Rapid eye movement sleep behavior disorder
* Major depressive disorder, schizophrenia, or other psychotic disorders, bipolar disorder, substance (including alcohol) related disorders
* Metal implants in the head (except dental), pacemaker, cochlear implants, or any other non-removable items that are contraindications to MRI
* Resides in hospital or moderate to high dependency continuous care facility
* History of swallowing difficulties
* Pregnant or breastfeeding
* Glucose-6-phosphate dehydrogenase deficiency
* History of significant hematological abnormality or current acute or chronic clinically significant abnormality
* Abnormal serum chemistry laboratory value at Screening deemed to be clinically relevant by the investigator
* Clinically significant cardiovascular disease or abnormal assessments
* Preexisting or current signs or symptoms of respiratory failure
* Concurrent acute or chronic clinically significant immunologic, hepatic, or endocrine disease (not adequately treated) and/or other unstable or major disease other than bvFTD
* Diagnosis of cancer within the past 2 years prior to Baseline (other than basal cell or squamous cell skin cancer or Stage 1 prostate cancer) unless treatment has resulted in complete freedom from disease for at least 2 years
* Prior intolerance or hypersensitivity to methylthioninium-containing drug, similar organic dyes, or any of the excipients
* Treatment currently or within 90 days before Baseline with any of the following medications (unless otherwise noted):

  * Tacrine
  * Amphetamine or dexamphetamine
  * Clozapine, olanzapine (and there is no intent to initiate therapy during the course of the study)
  * Carbamazepine, primidone
  * Drugs for which there is a warning or precaution in the labeling about methemoglobinemia at approved doses
* Current or prior participation in a clinical trial as follows:

  * Clinical trial of a product for cognition within 3 months of Screening (unless confirmed to have been randomized to placebo)
  * A clinical trial of a drug, biologic, device, or medical food in which the last dose/administration was received within 28 days prior to Baseline

Max Age: 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2013-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on Addenbrooke's Cognitive Examination - Revised (ACE-R) | 52 weeks
Change from Baseline on Functional Activities Questionnaire (FAQ) | 52 weeks
Change from Baseline on whole brain volume (assessed by brain MRI) | 52 weeks

SECONDARY OUTCOMES:
Change from Baseline on Unified Parkinson's Disease Rating Scale (UPDRS Parts II and III) | 52 weeks
Change from Baseline on Frontotemporal Dementia Rating Scale (FRS) | 52 weeks
Change from Baseline on Modified Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (modified ADCS-CGIC) | 52 weeks
Number of study participants who tolerate oral doses of TRx0237 as determined by safety parameter changes | 52 weeks
  Safety parameters included adverse events, vital signs, methemoglobin and oxygen saturation, physical and neurological examinations, laboratory tests (hematology, serum chemistry, and urinalysis), electrocardiograms, assessment of serotonin syndrome, brain magnetic resonance imaging (MRI) and potential for suicidal behavior and thoughts

OTHER OUTCOMES:
Early effect on modified ADCS-CGIC (change from Baseline) | 8 weeks
Change from Baseline on the rate of atrophy in frontal and temporal lobes as well as ventricular volume (assessed by brain MRI) | 52 weeks
Change from Baseline on Mini-Mental Status Examination (MMSE) | 52 weeks
Change from Baseline on Addenbrooke's Cognitive Examination-III (ACE-III) | 52 weeks
Determine the effect of TRx0237 in subjects with known genetic mutations associated with bvFTD | 52 weeks

CONTACTS AND LOCATIONS:
Locations (67):
- United States (24):
  - David Geffen School of Medicine at UCLA, UCLA Neurological Services, Los Angeles, California
  - The Shankle Clinic, Newport Beach, California
  - Memory and Aging Centre, San Francisco, California
  - Meridien Research, Brooksville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Compass Research, LLC, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Department of Neurology, Emory University, Atlanta, Georgia
  - Alexian Brothers Neurosciences Institute Clinical Research, Elk Grove Village, Illinois
  - Indiana University Department of Neurology, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Neurological Clinical Research Institute (NCRI) Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Department of Neurology, Rochester, Minnesota
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - Neurological Associates of Albany, P. C., Albany, New York
  - Integrative Clinical Trials LLC, Brooklyn, New York
  - UNC Department of Neurology, Physicians Office Building, Chapel Hill, North Carolina
  - University Hospitals Case Medical Center, Neurology Clinical Trials Unit, Cleveland, Ohio
  - Rivers Wellness and Research Institute, Oklahoma City, Oklahoma
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Hospital of the University of Pennsylvania, Department of Neurology, Philadelphia, Pennsylvania
  - PRA Health Sciences, Phase 2/3 Outpatient and CNS Clinic, Salt Lake City, Utah
  - The Memory Clinic, Bennington, Vermont
  - University of Virginia, Charlottesville, Virginia
- Australia (3):
  - Neuroscience Research Australia, Randwick, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - Neurodegenerative Disorders Research Pty Ltd, West Perth, Western Australia
- Canada (8):
  - Heritage Medical Research Clinic-University of Calgary, Calgary, Alberta
  - University of British Columbia Hospital, Clinic for Alzheimer Disease and Related Disorders, Vancouver, British Columbia
  - Vancouver Island Health Authority, Victoria, British Columbia
  - True North Clinical Research, Halifax, Nova Scotia
  - Geriatric Clinical Trials Group, Parkwood Institute, London, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - University Health Network, Toronto Western Hospital, Memory Clinic, Toronto, Ontario
  - McGill Centre for Studies in Aging, Alzheimer Disease Research Unit, Verdun, Quebec
- Croatia (2):
  - University Hospital Centre Zagreb, Zagreb
  - University Psychiatric Hospital Vrapče, Zagreb
- Germany (5):
  - Charité-Universitätsmedizin Berlin Klinik für Psychiatrie und Psychotherapie, Berlin
  - Memory Clinic, ECRC, Berlin
  - Universitätsklinikum Hamburg-Eppendorf Klinik für Psychiatrie und Psychotherapie, Hamburg
  - Klinik und Poliklinik für Psychiatrie und Psychotherapie der Technischen Universität München, München
  - Universitäts - und Rehabilitationskliniken Ulm, Neurologie, Ulm
- Italy (4):
  - Unità di Neuroimmagine e Epidemiologia Alzheimer, Brescia
  - Fondazione Universita' Gabriele D'Annunzio di Chieti, Chieti Scalo
  - Fondazione IRCCS Istituto Neurologico "Carlo Besta", Milan
  - Neurology I, Department of Neuroscience, University of Torino, Torino
- Netherlands (3):
  - Jeroen Bosch Ziekenhuis, afdeling geriatrie, 's-Hertogenbosch
  - Alzheimer Research Center Amsterdam, Amsterdam
  - Erasmus University Medical Center, Rotterdam
- Poland (2):
  - NZOZ Neuro-Kard Ilkowski i Partnerzy Spółka Partnerska, Poznan
  - Euromedis Sp. z o.o., Szczecin
- Psychomedical Consult, Bucharest, Romania
- National Neuroscience Institute Department of Neurology, Singapore, Singapore
- Spain (3):
  - Fundació ACE. Institut Català de Neurociències Aplicades, Barcelona
  - Ceuta University Hospital; Neurology, Ceuta
  - Hospital Viamed Montecanal, Neurology Department, Zaragoza
- United Kingdom (11):
  - NHS Grampian, OAP Directorate, Aberdeen
  - The Barberry Out-Patients Department, Birmingham
  - 2gether NHS foundation trust, Cheltenham
  - Kingsway Hospital, Derby
  - St Margaret's Hospital Mental Health Unit, Epping
  - Cognition Health Ltd., London
  - Imperial College Healthcare NHS Trust - Charing Cross Hospital, London
  - Dementia Research Center at Queens Square, London
  - Nuffield Department of Clinical Neurosciences, Oxford
  - Redwoods Centre, Shrewsbury
  - Wessex Neurological Centre, Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Pletnikova O, Sloane KL, Renton AE, Traynor BJ, Crain BJ, Reid T, Zu T, Ranum LP, Troncoso JC, Rabins PV, Onyike CU. Hippocampal sclerosis dementia with the C9ORF72 hexanucleotide repeat expansion. Neurobiol Aging. 2014 Oct;35(10):2419.e17-21. doi: 10.1016/j.neurobiolaging.2014.04.009. Epub 2014 Apr 18. PMID 24819148